CLINICAL TRIAL: NCT06767072
Title: Effectiveness of Tailored Multichannel Interventions on Weight Loss Among Adolescents: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Prince Sattam Bin Abdulaziz University (Other); Mansoura University (Other); British University In Egypt (Other); Port Said University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Ahmed Ahmed Elsheikh, Lecturer, Faculty of Nursing, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB0689
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-01

CONDITIONS: Obesity Prevention; Obesity; Overweight Adolescents; Overweight/Obesity, Adolescent; BMI; Behaviour Change; Health Promotion; Health Behavior, Risky
Keywords: digital intervention.; overweight, adolescents, tailored, health belief model, multichannel; face-to-face college meetings, telephone calls, WhatsApp text messages, and digital intervention.
MeSH Terms: conditions — Obesity; Overweight; Health Risk Behaviors

STUDY DESIGN:
Intervention Model Description: prospective, open label, barreled two groups. the study participants will be assigned randomly to intervention group or control group. the participants in the the intervention group will receive the tailored Multichannel Interventions, while the control group will receive two supportive session. the intervention group will not receive the tailored multichannel intervention.
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): The CG is provided general information on overweight and obesity, and general advice to manage their weight. these will be explained to them during two college visits. CG participants will not receive tailored multichannel interventions.
- Intervention Group (Experimental): the intervention group will receive the Tailored Multichannel interventions that will be designed by an interdisciplinary team including academic researchers from different specialties.
  The proposed intervention will be administered by 8 intervention nurses via multiple channels.
  The current intervention will be delivered using the various modes for 5 months
  Interventions: Behavioral: Tailored Multichannel interventions

INTERVENTIONS:
Behavioral: Tailored Multichannel interventions — To ensure the feasibility of the intervention, the intervention will be designed by an interdisciplinary team including academic researchers from different specialties (experts in the fields of community health, psychiatry health, and nutrition), as well as 3 research assistants.
  The designing process for each individual in the intervention group involved the following 4 subsequent steps: (1) intervention nurses assess HBM constructs, which are used to collect data on each unique perception regarding overweight(Saghafi-Asl et al., 2020). (2) data are reviewed, identified, and summarized by the interdisciplinary team; (3) the interdisciplinary team then creates an intervention plan based on the summarized needs and (4) the intervention plan will be shared with the participant to ensure collaboration.
  The intervention will adopt the strategies of the Diabetes Prevention Program (DDP) (The Diabetes Prevention Program (DPP), 1996).
  Arms: Intervention Group

SUMMARY:
overweight among adolescents is a public health issue. However, several weight loss interventions were developed and conducted for adolescents. These interventions are often not adequately tailored to the needs of this vulnerable target group. Besides, these interventions proposed one channel is adequate to deliver the message to adolescents.

The proposed study aims to evaluate the effectiveness of tailored multichannel interventions on weight loss among adolescents.

The proposed study is a prospective, cluster-randomized controlled trial. 279 adolescents will be recruited from 8 non-medical colleges in Mansoura University. The 8 colleges will be randomly assigned to 4 colleges for the tailored multichannel nursing intervention or 4 colleges as a control group. For intervention participants, the tailor-based intervention will be designed and guided by a health belief model and take into evidence-based recommendations. The intervention will be designed by a multidisciplinary team and will be administered by 8 nurses for 5 months, including five face-to-face school meetings, five school-based telephone calls, and five WhatsApp text messages. Control group participants will receive 2 non-tailored face-to-face sessions. The primary outcome is the mean difference in weight loss between groups. The proposed study hypothesizes that the participants who will receive tailored multichannel intervention will lose significantly more weight (Body Mass Index) compared with the control group. Secondary outcomes include a health belief model.

DETAILED DESCRIPTION:
Overweight and obesity and their related consequences are largely preventable and manageable. However, overweight is one of the most common health problems in the world. World Health Organization (WHO) reported that 12.5 % of people worldwide are overweight according to a survey of the global burden of diseases conducted in 2022. Furthermore, worldwide adult obesity has more than doubled since 1990, and adolescent obesity has quadrupled. WHO, 2024 reported that 390 million children and adolescents aged 5-19 years were overweight including 160 million who were living with obesity. Overweight and obesity are significantly correlated with an increased risk of several health disorders, such as cardiovascular disease, psychological disturbance, metabolic syndrome, type 2 diabetes, fatty liver disease, and premature death. Obesity also imposes enormous financial burdens on governments and individuals. Adolescence obesity is of particular concern as it has increased globally, and it could have adverse health impacts in adulthood.

Overall, the global prevalence of adolescent obesity is a growing public health concern, with significant physical and psychological consequences. Adolescence is a critical period where dietary habits and lifestyle behaviors are shaped, making it an ideal time for interventions aimed at promoting healthy weight management. Several preventive and treatment interventions have been conducted to enhance weight control among adolescents in different countries. However, the effectiveness of past interventions has shown inconsistent outcomes. Compliance with weight-loss treatments varies for a range of reasons, mainly related to the design and delivery of the interventions.

Systematic reviews reveal debate regarding how best to motivate adolescents to manage their ideal body weight. Empirical evidence shows that tailored interventions are often considered more effective than standardized interventions for reducing overweight among adolescents. Tailored interventions account for individual differences in lifestyle, preferences, perceptions about health and obesity, and self-efficacy. Previous studies have shown that these factors play important roles in the success of weight loss and maintenance programs. While standardized interventions can provide a solid foundation, tailoring strategies to individual needs often leads to more sustainable behavior changes and better health outcomes. Tailored interventions consider each adolescent's unique motivations, preferences, and challenges. This personalization can lead to greater engagement and adherence.

The literature suggests that interventions delivered through multiple channels-such as social media, face-to-face interactions, and telephone calls-are often more effective in addressing overweight and obesity among adolescents. Adolescents are highly engaged with digital platforms like social media, making it a natural channel of communication and providing daily reminders or motivation. Incorporating face-to-face interactions builds a personal connection and offers in-depth discussions, while telephone calls provide a direct and accessible line of communication.

ELIGIBILITY:
Inclusion Criteria:

* Students in the first and second grades of college whose body mass index (BMI) of 25 or higher at the baseline assessment will be eligible to participate in the study.

Exclusion Criteria:

* Students will be excluded if they have one of the following criteria.

  * Students who report a physical condition or chronic illness or impairment preventing them from being physically active
  * Students who have physical conditions that prevent them from losing excess body weight
  * Students who are on medication that causes weight gain
  * Students with a history of mental health disorders
  * Students participating in another weight loss program

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 279 (Actual)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
BMI | All data related to primary and secondary outcomes will be collected at baseline (T0) at 2 (T1) months, and 5 months (T2) after the start of intervention.
  Weight in kg and height in cm will be assessed. BMI will be measured, calculated, and interpreted based on WHO guidelines and using BMI charts. Overweight is considered when a BMI is 25 kg/m2 and Obesity is equivalent to a BMI of 30 kg/m2 or over (WHO, 2024).

SECONDARY OUTCOMES:
Health belief model construct | All data related to primary and secondary outcomes will be collected at baseline (T0) at 2 (T1) months, and 5 months (T2) after the start of intervention.
  The key constructs of the HBM include 89 statements.(Jones et al., 2015) (Albasheer et al., 2024). Each statement will be rated on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). 13 questions evaluated perceived severity on three subscales (emotional/mental, health, physical health/fitness, and social professional). 7 questions evaluated perceived susceptibility and consisted of two subscales (lifestyle and environmental). 14 questions dealt with perceived barriers, comprising three subscales (practical concerns, emotional/mental health, and awareness). 13 questions on perceived benefits included three subscales (emotional/mental health, physical health/fitness, and social/professional). The 12 questions on cues to action consisted of two subscales (internal and external cues to action). 18 questions assessed self-efficacy in dieting and included two subscales (habits, preferences and emotional/mental health). The 7 questions on self-efficacy in exerc

CONTACTS AND LOCATIONS:
Overall Officials: M A ELSHEIKH, PhD, Principal Investigator — Cairo University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the investigators intended to share all data as ICMJE policy. IPD will be shared after the completion of the study. Data repository platform will be decided later.